CLINICAL TRIAL: NCT04180137
Title: A Single-center Randomized Controlled Comparative Interventional Prospective Study for Management of Endothelial Dysfunction in Patients With Chronic Venous Insufficiency After Endovenous Surgical Procedure Combined With and Without Additional Pharmacotherapy.
Brief Title: Management of Endothelial Dysfunction in Patients With Chronic Venous Insufficiency After Endovenous Surgical Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NMSC-02-19
Record Dates: First submitted 2019-11-21; First posted 2019-11-27 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Venous Insufficiency of Leg; Venous Insufficiency (Chronic)(Peripheral); Endothelial Dysfunction
MeSH Terms: conditions — Venous Insufficiency | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical treatment with subsequent pharmacotherapy (Experimental)
  Interventions: Procedure: Endovenous laser ablation of great saphenous vein (GSV) and microphlebectomy of varicose veins; Drug: Pharmacotherapy
- Isolated surgical treatment (Other)
  Interventions: Procedure: Endovenous laser ablation of great saphenous vein (GSV) and microphlebectomy of varicose veins

INTERVENTIONS:
Procedure: Endovenous laser ablation of great saphenous vein (GSV) and microphlebectomy of varicose veins — Surgical treatment is performed as endovenous laser ablation of GSV and microphlebectomy of varicose branches according to a standard protocol:
  The intervention includes treatment of the pathological upright reflux and varicose veins. Ultrasound-guided GSV puncture at the upper third of the leg under local anesthesia. The light guide is inserted into the vein lumen and pushed through to the saphenofemoral junction. Under ultrasound guidance the light guide is positioned at v. epigastrica superficialis junction. Under ultrasound guidance tumescent anesthesia is produced around the GSV from puncture site up to the saphenofemoral junction. Laser coagulation (with radial light guide), linear energy density - 75 J/cm, automatic traction of the light guide at the speed 0.7 mm/sec. Varicose veins are resected through skin punctures using Varady hook 1-2 mm.
Drug: Pharmacotherapy — After surgical intervention the active treatment group will receive sulodexide 250 lipasemic units (LSU) bid for 30 days.
  Arms: Surgical treatment with subsequent pharmacotherapy

SUMMARY:
Endothelial dysfunction is assessed in patients with chronic venous insufficiency of lower limbs (grade C4 according to C - clinical manifestations, E - etiologic factors, A - anatomic distribution of disease, and P - underlying pathophysiologic findings (CEAP) classification) prior to and after endovenous surgical procedure, i.e. endovenous laser ablation of great saphenous vein, microphlebectomy of varicose branches. Two treatment groups (with and without additional pharmacotherapy) are compared.

DETAILED DESCRIPTION:
Each patient will be examined 4 times:

Visit 1 (day -1)

* collecting and documenting patients' complaints and medical history
* local examination
* ultrasound angiography of the lower limbs veins
* assessment of clinical grade according to CEAP classification

Visit 2 (day 0)

* assessment of venous disease severity according to Venous Clinical Severity Score (VCSS)
* assessment of quality of life with Chronic Venous Insufficiency Quality of Life Questionnaire (CIVIQ-20)
* assessment of clinical grade according to CEAP classification
* measurement of microcirculation in the operated limb by laser flowmetry using portable device (laser Doppler flowmetry (LDF) registration will be performed on leg anterior surface (lower third) for 10 minutes)
* assesment of blood laboratory parameters of endothelial dysfunction: homocysteine, von Willebrand factor, plasminogen activator inhibitor-1 (PAI-1), E-selectin, P-selectin, soluble intercellular adhesion molecule-1 (sICAM-1), soluble vascular endothelial cell adhesion molecule-1 (sVCAM-1)
* flow cytometry analysis of circulating cells expressing surface markers (clusters of differentiation (CD)): CD 45-, CD 34+, CD 146+, CD 31+, CD 105+ and CD 309+
* surgical treatment is performed as endovenous laser ablation of GSV and microphlebectomy of varicose branches according to a standard protocol
* patients' randomization (method of random numbers) into 2 treatment groups of 20 subjects each with sulodexide treatment (250 LSU bid for 30 day) for the active treatment group and without any additional pharmacotherapy for the control group

Visit 3 (day 4 after intervention)

- ultrasound angiography of the operated limb (evaluation of the venous ablation and examination of endothermal heat-induced thrombosis (EHIT))

Visit 4 (day 32 after intervention)

* collecting and documenting patients' complaints
* local examination
* ultrasound angiography of the lower limbs veins
* assessment of clinical grade according to CEAP classification
* assessment of venous disease severity according to VCSS
* assessment of quality of life with CIVIQ-20
* measurement of microcirculation in the operated limb by laser flowmetry using portable device
* assesment of blood laboratory parameters of endothelial dysfunction: homocysteine, von Willebrand factor, PAI-1, E-selectin, P-selectin, sICAM-1, sVCAM-1
* flow cytometry analysis of circulating cells expressing surface markers: CD 45-, CD 34+, CD 146+, CD 31+, CD 105+ and CD 309+

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-65 years inclusive.
* Diagnosis: varicose veins of lower limbs in the GSV territory.
* Maximum diameter of target vein (GSV) - 15 mm.
* Clinical grade C4 according to CEAP classification.
* Absence of chronic diseases or acute diseases requiring first-line treatment.

Exclusion/withdrawal Criteria:

* Conditions that limit patient's adherence to study procedures (dementia, neuropsychological disorders, substance and alcohol dependence, etc.).
* Participation in other clinical trials (or administration of investigational medicinal products) within 3 months prior to the study.
* Patient's withdrawal from the study.
* History of thrombosis of superficial and/or deep veins of lower limbs at enrollment into the study.
* Current anticoagulant and phlebotropic therapy.
* Comorbidities requiring first-line treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in circulating endothelial cells | baseline and 32 days after surgery
  Flow cytometry analysis of circulating cells expressing surface markers: CD 45-, CD 34+, CD 146+, CD 31+, CD 105+ and CD 309+

SECONDARY OUTCOMES:
Changes in microcirculation | baseline and 32 days after surgery
  Measurement of microcirculation of the operated limb by laser flowmetry using portable device equipped with laser Doppler flowmetry (LDF). LDF registration will be performed at leg anterior surface (lower third) for 10 minutes.
  The results of measurements will be automatically analyzed and fixed in single protocol which includes the following parameters:
  * Mean value of tissue blood perfusion.
  * Flux amplitude - standard deviation for oscillations of microcirculation values at given time interval.
  * Flux motion index.
  * Spectral analysis of blood flow oscillations with determination of oscillation amplitude at given frequency band, as well as determination of contribution of certain frequency bands into total power of biological rhythm spectrum.
  * Microvascular tone and intravascular resistance
  * Microvascular reactivity and functional reserve of the capillary bed with the help of functional tests.
Changes in quality of life | baseline and 32 days after surgery
  Quality of life assessed with CIVIQ-20. The 20-item questionnaire, which provides a global index and an outline of 4 quality-of-life dimensions-"pain" (4 items), "physical" (4 items), "psychological" (9 items), and "social" (3 items). Items on the CIVIQ-20 scale are scored from 1 to 5. A low score corresponds to greater patient comfort, high score represents worse life quality.
Changes in severity of disease | baseline and 32 days after surgery
  Severity of disease estimated by Venous Clinical Severity Score (VCSS). It is used to assess those with venous disease that that is complementary to the CEAP classification. The score includes 10 clinical parameters (pain, varicose veins, venous edema, skin hyperpigmentation, inflammation, induration, number of ulcers, durations of ulcers, size of ulcers, and compliance with compression therapy). Each item is graded from zero to three depending on severity (None = 0, Mild = 1, Moderate = 2, Severe = 3). The lower the score the less severity, the higher the score the more severity.
Changes in homocystein level | baseline and 32 days after surgery
  Assesment of blood homocysteine as a laboratory parameter of endothelial dysfunction.
Changes in von Willebrand factor level | baseline and 32 days after surgery
  Assesment of blood von Willebrand factor as a laboratory parameter of endothelial dysfunction.
Changes in PAI-1 level | baseline and 32 days after surgery
  Assesment of blood PAI-1 as a laboratory parameter of endothelial dysfunction.
Changes in E-selectin level | baseline and 32 days after surgery
  Assesment of blood E-selectin as a laboratory parameter of endothelial dysfunction.
Changes in P-selectin level | baseline and 32 days after surgery
  Assesment of blood P-selectin as a laboratory parameter of endothelial dysfunction.
Changes in sICAM-1 level | baseline and 32 days after surgery
  Assesment of blood sICAM-1 as a laboratory parameter of endothelial dysfunction.
Changes in sVCAM-1 level | baseline and 32 days after surgery
  Assesment of blood sVCAM-1 as a laboratory parameter of endothelial dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri M Stoyko, Prof, Principal Investigator — N.I. Pirogov National Medical and Surgical Center
Locations (1):
- N.I. Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 6 months after completion of the study
Access Criteria: upon request